CLINICAL TRIAL: NCT02737358
Title: Evaluating N-acetylcysteine as a Pharmacotherapy for Tobacco Use Disorder
Brief Title: N-acetylcysteine for Tobacco Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin McClure, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro 00052793; R34DA042228 (NIH)
Record Dates: First submitted 2016-03-14; First posted 2016-04-13 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Nicotine Dependence; Smoking
Keywords: nicotine; tobacco; smoking; cessation; N-acetylcysteine; NAC; pharmacotherapy; relapse; tobacco use disorder
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Recurrence | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo will be given to half of the study participants.
  Interventions: Other: Placebo
- N-Acetylcysteine (NAC) (Active Comparator): NAC will be given to half of the study participants. The dose of NAC will be 2400 mg per day (1200 mg taken twice per day as two 600 mg capsules)
  Interventions: Drug: N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — NAC or matched placebo will be given to study participants for 8 weeks.
  Other Names: NAC
  Arms: N-Acetylcysteine (NAC)
Other: Placebo — Matched placebo (2 capsules taken in the morning and evening) will be taken by study participants for eight weeks. All participants will receive brief smoking cessation counseling and support.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of administering N-Acetylcysteine (NAC) to assist in initial cessation and/or relapse prevention in adult cigarette smokers.

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of N-acetylcysteine (NAC) on initial cessation and relapse prevention in adult cigarette smokers. Specifically, this study has the following aims: Aim 1) Examine the efficacy of NAC, compared to placebo, in helping smokers achieve three days of continuous abstinence; Aim 2) Among those who maintain initial 3-day abstinence, examine the time to relapse over the 8-week intervention between NAC and placebo groups; Aim 3) Assess 7-day point prevalence abstinence at the 8-week end-of-treatment study visit in order to obtain effect sizes and estimates of variability to power a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Daily smoker for ≥6 months, smoking approximately ≥5 cigarettes per day on average in the past month or must meet the criteria for nicotine dependence
3. Be interested in quitting smoking (defined as a 2 or above on a 10-point Likert scale assessing readiness and interest in quitting (1=not at all ready/interested, 10=extremely ready/interested)
4. Willing to engage in a 3-day quit attempt as part of study procedures
5. Willing to abstain from cannabis use during study procedures (since inhaled cannabis will affect breath carbon monoxide readings).
6. If female, agreement to use birth control (any form) to avoid pregnancy during study procedures

Exclusion Criteria:

1. Any serious or unstable medical/psychiatric disorder (including severe substance use disorders, other than tobacco use disorder) in the past month that may interfere with study performance based on PI judgment
2. Current pregnancy or breastfeeding
3. Current use of medications with smoking cessation efficacy
4. Known hypersensitivity to NAC
5. Use of carbamazepine or nitroglycerin (or any other medication deemed to be hazardous if taken with NAC) within 14 days of study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tomko RL, Gray KM, Oppenheimer SR, Wahlquist AE, McClure EA. Using REDCap for ambulatory assessment: Implementation in a clinical trial for smoking cessation to augment in-person data collection. Am J Drug Alcohol Abuse. 2019;45(1):26-41. doi: 10.1080/00952990.2018.1437445. Epub 2018 Mar 7. PMID 29513609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult daily cigarette smokers were recruited from the community in Charleston, South Carolina (US).
Pre-assignment Details: Following screening, participants completed mobile daily diaries leading up to a Training visit. During this visit, participants were instructed on how to leave a carbon monoxide samples, upload videos, and loaned equipment to complete remote samples. Prior to randomization, 22 participants withdrew, were lost to follow-up or were discontinued.
Period: Overall Study
Arm/Group | Placebo | N-Acetylcysteine (NAC)
Started | 55 | 59
Completed | 46 | 44
Not Completed | 9 | 15
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | N-Acetylcysteine (NAC) | Total
Number analyzed (Participants) | 55 | 59 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 59 | 114
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (11.4) | 40.2 (12.2) | 42.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 27 | 29 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 49 | 57 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 21 | 33
  White | 38 | 36 | 74
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemically-verified Abstinence From Smoking on Days 1-3 of the Protocol.
Description: Abstinence will be measured through biochemical verification via breath carbon monoxide. Abstinence is defined as a 75% reduction in carbon monoxide values (parts per million) from smoking baseline levels.
Time Frame: Days 1-3 of the study protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | N-Acetylcysteine (NAC)
Number analyzed (Participants) | 55 | 59
Participants | 8 | 6

2. Secondary Outcome: Days to Relapse to Smoking Among Abstinent Participants
Description: Relapse to smoking will be measured through carbon monoxide-verified relapse at weekly study visits among those who abstained during the 3-day quit attempt. Relapse (return to smoking) will be defined as carbon monoxide values (in parts per million) that do not meet abstinence criteria (i.e., 75% reduction from baseline smoking levels).
Time Frame: Days 4-56 of the study protocol
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | N-Acetylcysteine (NAC)
Number analyzed (Participants) | 55 | 59
days | 17.0 (3.45) | 3.8 (1.35)

3. Secondary Outcome: Number of Participants With 7-day Point Prevalence Abstinence at the 8-week End-of-treatment Visit
Description: Seven day point prevalence abstinence will be measured through biochemical verification via breath carbon monoxide and urinary cotinine analysis. Abstinence is defined as a 75% reduction in carbon monoxide values (parts per million) from smoking baseline levels and a negative urine cotinine measure (<80 ng/mL).
Time Frame: Days 49-56
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | N-Acetylcysteine (NAC)
Number analyzed (Participants) | 46 | 44
Participants | 6 | 4

ADVERSE EVENTS:
Time Frame: 3 months (randomization to last post-treatment follow-up visit)
Description: Assessed and coded in MedDRA terminology by the medical clinician at each visit.
Arm/Group | Placebo | N-Acetylcysteine (NAC)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/59
Other Adverse Events (participants affected / at risk) | 32/55 | 33/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | N-Acetylcysteine (NAC) (N=59)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Hypertension (worsening) (Vascular disorders) | 2 (2) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain (Worsening) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermatitis Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Influenza Like Illness (Infections and infestations) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Malposition Teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Mood Swings (Psychiatric disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peri-umbilical Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Post Operative Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sprained Knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomachache (Gastrointestinal disorders) | 3 (3) | 3 (3)
Tachycarida (Cardiac disorders) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 12 (12) | 8 (8)
Vivid Dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT02737358/Prot_SAP_000.pdf